CLINICAL TRIAL: NCT05407844
Title: Community Health Worker Based Intervention to Improve Palliative Care
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00119097; 1R01CA252101-01A1 (NIH); 1R01MD016935-01 (NIH); IRB00283002 (Other: Johns Hopkins (old IRB #))
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Cancer; End Stage Cancer; Malignancy; Advanced Cancer
Keywords: palliative care; community health worker
MeSH Terms: conditions — Neoplasms | interventions — Community Health Workers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Standard cancer care
- Standard care + DeCIDE PC intervention (Experimental): Community health worker support and standard cancer care
  Interventions: Other: Community Health Worker (CHW) based palliative care

INTERVENTIONS:
Other: Community Health Worker (CHW) based palliative care — Those in the intervention group will receive support from a dedicated CHW trained in motivational interviewing, components of palliative care communication, and social determinants of health.
  Arms: Standard care + DeCIDE PC intervention

SUMMARY:
The study aims to find out if community health worker (CHW) support will improve palliative care outcomes in African American patients with advanced cancer, by comparing the quality of life of patients who are receiving standard care to those whose standard care is supplemented with CHW support.

DETAILED DESCRIPTION:
This research is being done to establish the effectiveness of a Community Health Worker based palliative care intervention among African American patients with advanced solid organ malignancies and their care givers.

The investigators' long-term goal is to reduce the research-to-practice gap in utilization of evidence-based palliative care (PC) in African Americans with advanced cancer. The objectives of this study are to establish the effectiveness of a CHW-based palliative care intervention and develop generalizable knowledge on how contextual factors influence implementation.

ELIGIBILITY:
Patient Inclusion Criteria:

* Self-identified African American patients with advanced (AJCC stage III or IV) solid organ malignancy
* >=18 years old
* English speaking
* Intact cognition and ability to provide informed consent

Patient Exclusion Criteria:

* Participants < 18 years of age
* Participants who are already receiving palliative care services

Caregiver Inclusion Criteria:

* Adult (>=18 years old) caregivers providing informal (unpaid) care to an eligible African American cancer patient (related or unrelated)
* English speaking
* Intact cognition and ability to provide informed consent

Caregiver Exclusion Criteria:

* Participants < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who completed Advance Directives | 6 months after enrollment
  Advanced care planning

SECONDARY OUTCOMES:
Functional Assessment of Chronic Illness Therapy-Palliative Subscale (FACIT-PAL) score | 6 months after enrollment
  Quality of Life; Score range: 0-184 [per scoring document, for total score] Higher scores signify better quality of life
Number of participants who utilize hospice care | 6 months after enrollment
  Hospice care utilization within 14 days of death (Yes/No)
Goals of care as assessed by Quality of communication (QOC) scale | 6 months after enrollment
  Goals of Care; Score range: 0-10 [scored 0-10 for each of 19 components] Higher scores signify: higher quality communication with physician
Symptom Intensity as assessed by the Edmonton Symptom Assessment Score (ESAS) | 6 months after enrollment
  Symptom; Score range: 0-10 [scored 0-10 for 10 components] Higher scores signify: higher intensity of cancer symptoms (worse symptoms)
Depression as assessed by the Center for Epidemiologic Studies Depression Scale (CES-D) | 6 months after enrollment
  Symptom; The score is the sum of the 20 questions. Possible range is 0-60. A score of 16 points or more is considered depressed.
Quality of life assessed by the 5-Level EuroQol 5-Dimensional (EQ-5D-5L) | 6 months after enrollment
  it assesses five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a visual analogue scale (VAS). Each dimension has five levels ranging from 1 (no problem) to 5 (extreme problem). Score range 0 to 100, higher score indicates better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Fabian M Johnston, MD, MHS, Principal Investigator — Johns Hopkins School of Medicine; Aarti Mathur, MD, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - TidalHealth Peninsula Regional, Inc., Salisbury, Maryland
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnston FM, Neiman JH, Parmley LE, Conca-Cheng A, Freund KM, Concannon TW, Smith TJ, Cooper LA. Stakeholder Perspectives on the Use of Community Health Workers To Improve Palliative Care Use by African Americans with Cancer. J Palliat Med. 2019 Mar;22(3):302-306. doi: 10.1089/jpm.2018.0366. Epub 2018 Nov 2. PMID 30388060
- [Derived] Monton O, Drabo EF, Masroor T, Fuller S, Woods AP, Siddiqi A, Malone TB, Johnston FM. Economic evaluation of a hybrid type 1 effectiveness-implementation trial comparing a community health worker palliative care intervention to enhanced standard of care in African American patients across four cancer centres in the USA: a study protocol. BMJ Open. 2025 Nov 4;15(11):e096402. doi: 10.1136/bmjopen-2024-096402. PMID 41193212
- [Derived] Siddiqi A, Monton O, Woods A, Masroor T, Fuller S, Owczarzak J, Yenokyan G, Cooper LA, Freund KM, Smith TJ, Kutner JS, Colborn KL, Joyner R, Elk R, Johnston FM. Dissemination and Implementation of a Community Health Worker Intervention for Disparities in Palliative Care (DeCIDE PC): a study protocol for a hybrid type 1 randomized controlled trial. BMC Palliat Care. 2023 Sep 18;22(1):139. doi: 10.1186/s12904-023-01250-0. PMID 37718442